CLINICAL TRIAL: NCT02625038
Title: CT-based Evaluation of the Intraoperative Implementation Accuracy of 3D-planned Osteotomies of the Hand and Forearm Performed With Patient-specific Instruments
Brief Title: Evaluation of the Intraoperative Accuracy of 3D-planned and Guided Osteotomies of the Hand and Forearm
Acronym: CARDFOREARM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-MD-0016
Record Dates: First submitted 2015-11-27; First posted 2015-12-09 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Posttraumatic or Congenital Bone Deformity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interventional (Experimental): 3D-planned osteotomies with patient-specific guides
  Interventions: Device: EUDAMED CIV-14-03-011940

INTERVENTIONS:
Device: EUDAMED CIV-14-03-011940

SUMMARY:
Target of the study is to evaluate the reduction accuracy of 3D computer-planned osteotomies that are performed with patient-specific instruments.

Due to the higher accuracy achieved it is expected that complaints can be resolved or effectively revealed. The Research hypothesis to prove is "The medical product permits the surgical reduction of deformed bones of the hand and forearm (radius, ulna, distal humerus, carpal, metacarpal, and finger bones) by corrective osteotomy within an accuracy of 2 mm and 2º. Secondary outcome is an assessment of the surgical outcome using the "Disabilities of the Arm, Shoulder and Hand" (DASH) and the "Patient related wrist Evaluation" (PRWE) scores.

ELIGIBILITY:
Inclusion criteria

* Posttraumatic or congenital bone deformity or pseudoarthrosis in the field of hand Surgery requiring correction by corrective osteotomy
* Clinical indication for a computer tomography scan of the forearms
* > 18 years old
* written informed consent

Exclusion criteria

* pregnant or nursing women
* other clinical significant accompanying symptoms (Tumor, infection)
* non-compliance of the patient to follow the clinical study protocol, drug or alcohol abuse
* Participation in a different clinical trial within the last 30 days before inclusion or during the study

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-09; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
3D difference between preoperative plan and surgery | 42 month
  For each reduced fragment the 3D difference in all 6 degrees of freedom (3xrotation, 3xtranslation) is quantified by comparing pre- and postoperative CT.

SECONDARY OUTCOMES:
Surgical Outcome | 42 month
  The surgical outcome is assessed by comparing DASH- and PRWE-scores pre- and postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Schweizer, Prof., Principal Investigator — University of Zurich
Locations (1):
- University Hospital Balgrist, Zurich, Switzerland